CLINICAL TRIAL: NCT06793033
Title: A Randomized Controlled Study of the NEURESCUE Device as an Adjunct to Advanced Cardiac Life Support
Acronym: ARISE RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: neurescue (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARISE RCT
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Cardiac Arrest (CA); Cardiopulmonary Arrest
MeSH Terms: conditions — Heart Arrest | interventions — Advanced Cardiac Life Support

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Control) (Active Comparator): Enrolled subjects randomized into Arm 1 will receive ACLS treatment.
  Interventions: Procedure: Advanced Cardiac Life Support (ACLS)
- Arm 2 (Intervention) (Experimental): Enrolled subjects randomized into Arm 2 will receive ACLS treatment combined with ABO.
  Interventions: Procedure: Advanced Cardiac Life Support (ACLS); Device: Aortic balloon occlusion (ABO)

INTERVENTIONS:
Procedure: Advanced Cardiac Life Support (ACLS) — Standard of care Advanced Cardiac Life Support (ACLS) consists of cardiopulmonary resuscitation (CPR), airway management, ventilation and defibrillation.
Device: Aortic balloon occlusion (ABO) — Aortic balloon occlusion (ABO) is a technique that diverts blood ﬂow towards the coronary and cerebral circulation. ABO is investigated as an adjunct to the treatment of cardiac arrest.
  In this study ABO is performed using the NEURESCUE Catheter, which is inserted through an introducer in the femoral artery, and thereby inserted into the aorta during uninterrupted Advanced Cardiac Life Support (ACLS). The balloon is then temporarily inflated as an adjunct to the treatment of cardiac arrest.
  Arms: Arm 2 (Intervention)

SUMMARY:
The NEURESCUE device is the first intelligent balloon catheter for aortic balloon occlusion (ABO), an emergency technique that supercharges blood flow to the heart and brain within one minute from deployment.

The catheter-based device is delivered via the femoral artery, temporarily inflating a soft balloon in the descending to redirect blood flow towards the upper body.

The purpose of this study is to compare the clinical safety and performance of Advanced Cardiovascular Life Support (ACLS) versus ACLS in combination with Aortic Balloon Occlusion (ABO) using the NEURESCUE device in subjects with cardiac arrest.

DETAILED DESCRIPTION:
Subjects will be randomized into two arms: ACLS treatment or ACLS + ABO treatment. Those in the ACLS treatment arm will receive standard of care treatment for cardiac arrest, while those in Arm 2 will receive ACLS in combination with ABO.

The NEURESCUE device is an aortic balloon catheter designed to temporarily occlude the aorta. During the treatment, the NEURESCUE Catheter will be placed in the descending aorta and be connected to the NEURESCUE Assistant. The NEURESCUE Assistant facilitates pressure-regulated inflation and deflation of the balloon.

Throughout the treatment, cardiac rhythm and return of spontaneous circulation (ROSC) will be monitored.

The subject will be monitored for a total of 4 visits, where a 90-days follow-up will account for the last visit.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤80 years
* Witnessed arrest
* CPR initiated within 7 min of arrest
* CPR time less than 40 min at enrollment
* Non-shockable rhythm

Exclusion Criteria:

* Traumatic cardiac arrest
* Known pregnancy
* Known terminal disease
* Known do-not-attempt-CPR order
* Known opposition to study participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Resuscitation | Measured from 10 minutes after randomization to 70 minutes after randomization
  Subject achieving shockable rhythm or ROSC

SECONDARY OUTCOMES:
Epinephrine | Measured from 10 minutes after randomization to 70 minutes after randomization
  Dosage of epinephrine administered during resuscitation
Procedures | Measured from 10 minutes after randomization to 90 days post cardiac arrest
  Need for any invasive procedures, e.g. surgery, extracorporeal membrane oxygenation (ECMO) or percutaneous coronary intervention (PCI)
(S)A(D)E | Measured from randomization to 90 days post cardiac arrest
  All Anticipated (S)AEs/(S)ADEs and Unanticipated (S)AEs/(S)ADEs
CPC score | Measured at dischage or at 7 days post cardiac arrest, and 90 days post cardiac arrest
  Cerebral Performance Category (CPC) is a five-point scale used to categorize the neurological outcome after cardiac arrest
EQ-5D | Measured 90 days post cardiac arrest
  EQ-5D is a standardized measure of quality of life
Survival | Measured at dischage or at 7 days post cardiac arrest, and 90 days post cardiac arrest
  Survival at discharge or 7 day post cardiac arrest (whichever comes first), and survival at 90 days post cardiac arrest

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Charité - Universitätsklinikum Berlin, Berlin
  - University Hospital Heidelberg, Heidelberg

IPD SHARING:
Plan to Share IPD: No
Individual request